CLINICAL TRIAL: NCT04748718
Title: Serial Movement Assessment in Athletes Who Perform Injury Prevention Training
Brief Title: Serial Movement Assessment in Collegiate Athletes Who Perform Injury Prevention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Vermont University (Other)
Responsible Party: Principal Investigator, Eleanor Beltz, Assistant Professor, Northern Vermont University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Beltz FAW2122 NMC PTP
Record Dates: First submitted 2021-01-31; First posted 2021-02-10 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Injury Leg; Injury, Knee; Injury;Sports; Injury, Ankle
Keywords: sport injury; injury prevention; neuromuscular control
MeSH Terms: conditions — Leg Injuries; Knee Injuries; Athletic Injuries; Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injury Prevention Arm (Experimental): exercise-based neuromuscular training injury prevention program
  Interventions: Other: Exercise-based injury prevention program

INTERVENTIONS:
Other: Exercise-based injury prevention program — ~10-minute, 4+ times/week exercise-based injury prevention program. Includes flexibility, strengthening, balance, agility and plyometric exercises.

SUMMARY:
Athletic injury can result in decreased athletic performance or removal from sport participation. There may also be psychological and financial impacts of athletic injury. Additionally, there can be long-term consequences, such as increased risk of subsequent injury or arthritis. Therefore, determining ways to prevent athletic injury from occurring is critical. Movement quality during sport is related to injury risk. Athletes who move poorly are generally at increased risk of injury compared to athletes who move well. Movement quality can be improved through exercise-based injury prevention training, thereby decreasing injury risk. This purposed of this study is to evaluate movement quality multiple times over the course of an athletic season in collegiate athletes who perform injury prevention training. The hypothesis is that movement quality will improve over the course of an athletic season.

DETAILED DESCRIPTION:
Neuromuscular control, or quality of movement, during sport is related to injury risk. Athletes who move poorly are generally at increased risk of injury compared to athletes who move well. Neuromuscular control can be improved through exercise-based injury prevention training (called preventive training programs, or PTPs), thereby decreasing injury risk. Neuromuscular control is dynamic and therefore should be evaluated regularly; however, no study has serially evaluated neuromuscular control in athletes who perform PTPs. The overall objective of the proposed study is to longitudinally evaluate multiple aspects of neuromuscular control (i.e., movement quality, balance) across several time points during a single athletic season in collegiate athletes who perform PTPs. Therefore, two specific aims are proposed: Specific Aim 1: Evaluate neuromuscular control at multiple time points during an athletic season in collegiate athletes who perform PTPs. Specific Aim 2: Evaluate multiple measures of neuromuscular control over the course of an athletic season in collegiate athletes who perform PTPs. A field-based, experimental, cohort study will be used to address both specific aims. Subjects will be recruited from NCAA-Division III men's and women's soccer, volleyball and basketball teams. Neuromuscular control will be assessed four times during the athletic season using the Landing Error Scoring System (LESS), the Balance Error Scoring System (BESS), and the Star Excursion Balance Test (SEBT). The LESS evaluates movement quality, while the BESS and the SEBT evaluate static and dynamic balance, respectively. Subjects will perform PTPs for about 10 minutes/day, at least 4 days/week.

ELIGIBILITY:
Inclusion Criteria:

* National Collegiate Athletics Association (NCAA) Division III Athlete
* Coach and athletic trainer elect to receive injury prevention services
* Ages 18-24

Exclusion Criteria:

-Does not participate on NCAA Division III Athletic Team

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Beltz, PhD, ATC, Principal Investigator — Northern Vermont University
Locations (1):
- Northern Vermont University, Johnson, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injury Prevention Arm
Started | 62
Completed | 12
Not Completed | 50
Not completed — Lost to Follow-up | 50

BASELINE CHARACTERISTICS:
Arm/Group | Injury Prevention Arm
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
height [Mean (Standard Deviation); unit: cm] | 180.3 (13.3)
mass [Mean (Standard Deviation); unit: kg] | 77.5 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Landing Error Scoring System (LESS) Score
Description: number of errors; scale is 0-17; lower score indicates better outcome
Time Frame: assessing change over 3 timepoints: baseline (week 0), midseason (weeks 4-6), end-of-season (weeks 10-12)
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Injury Prevention Arm
Number analyzed (Participants) | 12
errors
  baseline | 6 (1.8)
  midseason | 5.8 (1.2)
  end-of-season | 5.2 (1.6)

2. Primary Outcome: Balance Error Scoring System (BESS) Score
Description: number of errors; scale is 0-60; higher score indicates worse outcome
Time Frame: assessing change over 3 timepoints: baseline (week 0), midseason (weeks 4-6), end-of-season (weeks 10-12)
Population: complete data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Injury Prevention Arm
Number analyzed (Participants) | 12
errors
  baseline | 28.6 (5.9)
  midseason | 22.5 (10.3)
  end-of-season | 25.9 (7.3)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 7 months
Arm/Group | Injury Prevention Arm
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04748718/Prot_SAP_000.pdf